CLINICAL TRIAL: NCT06347835
Title: Biomarker Identification and Nutritional Intervention of Primary Sarcopenia Based on Gut-muscle Axis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yu Kang, MD, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gut-Intervention-SAR-2024
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Gut-muscle Axis; Biomarker; Gut microbiota; Intervention
MeSH Terms: conditions — Sarcopenia | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- symbiotic and whey protein intervention (Experimental): This group received dietary guidance, symbiotic and whey protein intervention for 12 weeks
  Interventions: Dietary Supplement: symbiotic; Dietary Supplement: whey protein
- whey protein intervention (Experimental): This group received dietary guidance and whey protein intervention for 12 weeks
  Interventions: Dietary Supplement: whey protein; Dietary Supplement: symbiotic placebo
- control (Placebo Comparator): This group received dietary guidance and maltodextrin for 12 weeks
  Interventions: Dietary Supplement: symbiotic placebo; Dietary Supplement: whey protein placebo

INTERVENTIONS:
Dietary Supplement: symbiotic — The intervention is made up of multiple probiotics and prebiotics (20g/d) and dietary pattern modification.
  Arms: symbiotic and whey protein intervention
Dietary Supplement: whey protein — The intervention is made up of whey protein supplements (20g/d) and dietary pattern modification.
  Arms: symbiotic and whey protein intervention; whey protein intervention
Dietary Supplement: symbiotic placebo — The intervention is made up of maltodextrin (20g/d) and dietary pattern modification.
  Arms: control; whey protein intervention
Dietary Supplement: whey protein placebo — The intervention is made up of maltodextrin (20g/d) and dietary pattern modification.
  Arms: control

SUMMARY:
The loss of skeletal muscle mass and function usually occurs with aging, known as primary sarcopenia. Sarcopenia has a prevalence of 11.6% among the elderly population in China and is closely associated with increased risks of falls, disability, and mortality. Currently, there is a lack of definition criteria for sarcopenia based on biomarkers. The Gut-Muscle Axis hypothesis suggests a complex interplay between gut microbiota and skeletal muscle. Nutritional intervention targeting the gut microbiota potentially plays a significant role in muscle regeneration. Therefore, this study aims to explore the effects of symbiotic and whey protein on muscle, gut microbiota, and clinical outcomes among sarcopenia patients, to provide a reference for further diagnosis and treatment of sarcopenia.

DETAILED DESCRIPTION:
This study will last 12 weeks. For the duration of the study, an anticipated total of 120 participants will be randomly assigned to three groups. During the study visits, questionnaires, blood and stool collection, and functional testing will occur. Intention-to-treat analysis (ITT) and per-protocol analysis (PP) will be conducted in statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 and older
2. Can cooperate with the measurement and questionnaire survey
3. Meets Asian Working Group for Sarcopenia (AWGS) 2019 diagnostic criteria for sarcopenia
4. Obtain informed consent to participate in this study

Exclusion Criteria:

1. Severe complications
2. Suffers from neuromuscular related diseases
3. Immobility
4. Have taken antibiotics, probiotics and other medications that may affect the gut microbiota in the last 6 weeks
5. Implants of electronic devices or metal objects in the body

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of Appendicular skeletal muscle mass index at 12 weeks | 12 weeks
  Defined as muscle mass (Unit: kg/m2)
Change from Baseline of grip strength at 12 weeks | 12 weeks
  Defined as muscle strength (Unit: kg)

SECONDARY OUTCOMES:
Change from Baseline of Short Physical Performance Battery score at 12 weeks | 12 weeks
  Measured by Short Physical Performance Battery (0-12) with higher scores meaning better physical performance.
Change from Baseline of gait speed at 12 weeks | 12 weeks
  Defined as gait speed (Unit: m/s)
Change from Baseline of gut microbiota composition at 12 weeks | 12 weeks
  The stool samples of participants before and after intervention will be collected and analyzed by 16S ribosomal RNA (rRNA).
Change from Baseline of inflammation status at 12 weeks | 12 weeks
  Inflammation status will be represented by Interleukin-6 (IL-6), IL-8, IL-10 and Tumour necrosis factor alpha (TNF-α).
Change from Baseline of microbiota-derived metabolites at 12 weeks | 12 weeks
  Microbiota-derived metabolites includes short-chain fatty acids, amino acid metabolites and secondary bile acids.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No